CLINICAL TRIAL: NCT06931613
Title: Autologous Hematopoietic Stem Cell Transplantation in Pediatric Relapsed or Refractory Hodgkin Lymphoma After Nivolumab Treatment With or Without Bendamustine
Brief Title: Autologous Hematopoietic Stem Cell Transplantation in Pediatric Relapsed or Refractory Hodgkin Lymphoma After Nivolumab Treatment
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Principal Investigator, Ivan S Moiseev, Professor, RM Gorbacheva Research Institute at First Pavlov State Medical University of St. Petersburg Russia, St. Petersburg State Pavlov Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 34/19-н
Record Dates: First submitted 2025-04-09; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Relapsed or Refractory Hodgkin Lymphoma; Children; Nivolumab; Autologous Haemopoietic Stem Cell Transplant
MeSH Terms: conditions — Recurrence; Hodgkin Disease | interventions — Nivolumab; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- The only ARM consists of nivolumab with or without bendamustine prior to auto-HSCT (Experimental)
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab with or without bendamustine is administered to children prior to auto-HSCT
  Other Names: bendamustine; autologous hematopoietic stem cell transplantation

SUMMARY:
Children with relapsed or refractory Hodgkin lymphoma receive 3-6 cycles of nivolumab monotherapy. In case of achieving complete response (CR) auto-HSCT is performed. In the absence of CR, 3-6 additional cycles of nivolumab with bendamustine are administered. If complete or partial response is achieved, auto-HSCT is performed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Hodgkin lymphoma established on the basis of histological and immunohistochemical studies
* Confirmation of relapsed of refractory Hodgkin lymphoma based on histological and immunohistochemical studies or based on imaging methods (PET/CT and/or CT).
* Number of previous lines of therapy >2
* Karnofsky index ≥60%
* availability of signed informed consent -

Exclusion Criteria:

* Number of previous lines of therapy ≤ 2
* Karnofsky index < 60
* Intolerance to drugs used in the study
* Presence of a second tumor
* Pregnancy or lactation
* Participation in another study within six months
* Presence of concomitant severe disease
* Presence of HIV and/or viral hepatitis (B or C)

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Event free survival | 5-year

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - N. N. Blokhin Russian Cancer Research Center, Moscow, Russia, Moscow
  - Pavlov University, RM Gorbacheva Research Institute, Saint Petersburg